CLINICAL TRIAL: NCT06103240
Title: Changes in the Gut Microbiota Composition of Healthy Young Volunteers After Administration of Lacticaseibacillus Rhamnosus LRa05: A Placebo-controlled Study
Brief Title: A Probiotic That Improve Intestinal Flora
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wecare Probiotics Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: WK2023004
Record Dates: First submitted 2023-10-21; First posted 2023-10-26 (Actual); Last update posted 2023-10-26 (Actual); Status verified 2023-10

CONDITIONS: Intestinal Flora

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotic group (Active Comparator): Bacterial count：100 billion CFUs Take one sachet per day for 4 weeks.
  Interventions: Other: Lacticaseibacillus rhamnosus LRa05
- Placebo group (Placebo Comparator): maltodextrin
  Interventions: Other: Lacticaseibacillus rhamnosus LRa05

INTERVENTIONS:
Other: Lacticaseibacillus rhamnosus LRa05 — Bacterial count:100 billion CFUs Take one sachet per day for 4 weeks.

SUMMARY:
Purpose: to verify the physiological properties of Lactobacillus rhamnosus LRa05.

Bacterial count:100 billion Test Objective: to test and collect the changes of intestinal flora before and after the daily use of LRa05 product.

DETAILED DESCRIPTION:
In order to validate the physiological properties of the 100 billion probiotic Lactobacillus rhamnosus LRa05 product and to gather sufficient evidence to test the changes in the intestinal flora before and after the daily use of the probiotic product, the test was conducted on 110 college students aged 18-25 years.

The primary outcome was to investigate the increase in the diversity of the gut flora and the increase in the peak levels of beneficial bacteria in the gut, and the secondary outcome was to investigate whether there was a significant improvement in the PSQI Pittsburgh Sleep Quality Index and the ISI Insomnia Severity Index.

ELIGIBILITY:
Inclusion Criteria:

1. PSQI Pittsburgh Sleep Quality Index scale score >6 and <18
2. ISI Insomnia Severity Index scale score >8 and <23

Exclusion Criteria:

1. People who have been diagnosed with diabetes or have high blood sugar are not recommended to participate in the test;
2. people whose daily diet is too light or too oily are not recommended to participate in the test; people with special dietary structure (e.g. ketogenic diet, etc.) caused by weight loss or other reasons, such as muscle gain and fat loss, are not recommended to participate in the test;
3. others with special conditions are not recommended to participate, such as those who are allergic to probiotic products;
4. pregnant women, lactating women and people under 19 and over 45 years old should not experiment;
5. people with unhealthy stomach and intestines are not recommended to participate in the test;
6. people with low body fat and BMI <23 are not recommended to participate in the test.

Ages: 19 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 110 (Actual)
Dates: Start 2022-04-20 (Actual); Primary Completion 2022-04-25 (Actual); Study Completion 2022-06-11 (Actual)

PRIMARY OUTCOMES:
intestinal flora test | 4 weeks
  Subjects took a packet of probiotics every day. Before taking probiotics, two weeks after taking probiotics, and after taking probiotics, fecal samples were collected, and fecal 16s rRNA was extracted using a DNA kit.

CONTACTS AND LOCATIONS:
Locations (1):
- Henan University of Technology, Zhengzhou, Henan, China

IPD SHARING:
Plan to Share IPD: No